CLINICAL TRIAL: NCT04220957
Title: Comparison Between Digital and Conventional Impression Techniques in Children: a Crossover Randomized Controlled Trial
Brief Title: Digital Versus Conventional Impression Techniques in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Lorenzo Franchi, Associate Professsor, University of Florence
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: LF8
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Dental Impression Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Impression Technique (Experimental): Impression with an intraoral scanner (TRIOS 3, 3Shape, Denmark)
  Interventions: Other: Digital Impression Technique
- Conventional Impression Technique (Active Comparator): Conventional impression with alginate (Orthoprint, Zhermack)
  Interventions: Other: Conventional Impression Technique

INTERVENTIONS:
Other: Digital Impression Technique — Digital impressions of both arches will be taken by using an intraoral scanner (Trios 3, 3Shape, Denmark) by adhering to the scanning pattern recommended by the company for routine diagnosis and recording.
  Arms: Digital Impression Technique
Other: Conventional Impression Technique — Conventional Impression Technique of both arches will be taken with alginate (Orthoprint, Zhermack) on conventional stainless steel impression trays.
  Arms: Conventional Impression Technique

SUMMARY:
The impression is a necessary step for the orthodontic diagnosis. Digital impression has recently been introduced by means of intraoral optical scanners. To date, few studies have compared the conventional alginate impression with the digital impression with intraoral scanners. These studies have shown that digital impression could have some advantages in terms of satisfaction and less discomfort for the pediatric patient. Only one study is randomized and has analyzed patients between 10 and 17 years of age. There are, therefore, no randomized trials for patients under 10 years of age.

The objective of the study is to compare the conventional alginate impression with the digital impression of both dental arches in orthodontic patients between 6 and 10 years of age with a randomized crossover design. In particular, the preference, comfort, impression taking time and other subjective aspects will be analyzed. This is a monocentric, controlled, superiority, randomized, crossover, open study.

Inclusion criteria:

- Orthodontic patients between 6 and 10 years of age.

Exclusion criteria:

* Noncompliant patients
* patients with syndromes or systemic diseases
* patients suffering from cleft lip and palate. The patient will be asked which of the 2 dental arch impression procedures they prefer. In addition, patients will be provided with a questionnaire including VAS (Visual Analogue Scale) for comfort, pain, gag reflex and breathing difficulty. The VAS will consist of scales from 0 to 10.

As for the calculation of the sample size, this has been done by considering a null hypothesis for a proportion of 50% in the preference between the two treatments and an alternative hypothesis of 80%. For alpha set at 0.05, a power of 80% and a dropout rate of 10%, 24 patients are required.

Descriptive statistics will be performed for all variables (frequency and percentage for qualitative variables and mean and standard deviation for quantitative variables). For the primary endpoint variable, impression procedure preference, the test will be performed for one proportion and the 95% confidence interval will be calculated using the Clopper-Pearson method.

With regard to the secondary endpoint variables, duration of the procedure, comfort, pain, gag reflex, breathing difficulty, the 2 procedures will be compared with the t-test for paired data.

An Intention-To-Treat analysis will be performed. In case more than 5 deviations from the protocol will occur, a sensitivity analysis will also be performed per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients between 6 and 10 years of age.

Exclusion Criteria:

* Noncompliant patients
* patients with syndromes or systemic diseases
* patients suffering from cleft lip and palate.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Patient's preference for either digital or conventional impression techniques | 30 minutes
  The patient will be asked "If you had to take another impression which one of the 2 impression techniques would you prefer?" The patient will mark on a sheet of paper which one of the 2 impression techniques he/she prefers.

SECONDARY OUTCOMES:
Comfort during impression taking | 15 minutes
  VAS (Visual Analogue Scale) from 0 to 10 with 0 corresponding to "very uncomfortable" and 10 corresponding to "maximum comfort"
Pain during impression taking | 15 minutes
  VAS (Visual Analogue Scale) from 0 to 10 with 0 corresponding to "no pain" and 10 corresponding to "very painful"
Gag reflex during impression taking | 15 minutes
  VAS (Visual Analogue Scale) from 0 to 10 with 0 corresponding to "no gag reflex" and 10 corresponding to "vomiting"
Respiratory difficulty | 15 minutes
  VAS (Visual Analogue Scale) from 0 to 10 with 0 corresponding to "no respiratory difficulty" and 10 corresponding to "maximum respiratory difficulty"
Duration of the impression procedure | 15 minutes
  Time recorded in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- SOD Odontostomatologia, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bosoni C, Nieri M, Franceschi D, Souki BQ, Franchi L, Giuntini V. Comparison between digital and conventional impression techniques in children on preference, time and comfort: A crossover randomized controlled trial. Orthod Craniofac Res. 2023 Nov;26(4):585-590. doi: 10.1111/ocr.12648. Epub 2023 Mar 20. PMID 36891891